CLINICAL TRIAL: NCT05421884
Title: Impact of Five Love Languages on Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jennifer Hoang, Student Primary Investigator, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002262
Record Dates: First submitted 2022-02-25; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer Patient and their significant other (Experimental): The intervention will implemented in all cancer patients and their significant others
  Interventions: Behavioral: 5 Love Languages

INTERVENTIONS:
Behavioral: 5 Love Languages — Emotional support will be given through utilizing the patient/partners specific Love Language (physical touch, words of affirmation, gifts, quality time, and acts of service).

SUMMARY:
The objective of this study is to evaluate the effectiveness of an intervention utilizing the Five Love Languages on quality of life (pain, depression, and anxiety) of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer with a significant other who attend a Texas Oncology couples support group will serve as the study population

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 weeks
  Pain will be measured through the MD Anderson Cancer Center Brief Pain Inventory and improvement will be measured by change in pain scale score (ranging from 0=no pain to 10= pain as bad as you can imagine) from pre to post survey.
Depression | 6 weeks
  Depression will be measured through the Patient Health Questionnaire (PHQ-9) scoring from 0 being not at all to 3 nearly every day of depression symptoms and improvement will be measured in by change in total scoring.
Anxiety | 6 weeks
  Anxiety will be measured through the Generalized Anxiety Disorder 7-item (GAD-7) scoring from 0 being not at all to 3 nearly every day of anxiety symptoms and improvement will be measured in by change in total scoring.

SECONDARY OUTCOMES:
Relationship Quality | 6 weeks
  This research study is also expected to measure improvement in the relationship of the cancer patient with their significant other. This improvement in relationship will be measured through the Funk and Rogge Couples Satisfaction Index which contains various scales from 0-6 or 0-5 with lowest satisfaction being 0 and highest being 5/6 and improvement will be measured in change in score from pre to post survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Oncology, Fort Worth, Texas, United States